CLINICAL TRIAL: NCT07352241
Title: Effect of the Injectable Platelet-rich Fibrin on the Orthodontically Induced Apical Root Resorption Following Non-extraction-based Orthodontic Treatment in Adults: A Randomized Controlled Clinical Trial.
Brief Title: Repeated Injections of i-PRF for Decreasing Root Resorption After the Orthodontic Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-1-2026
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Crowding of Anterior Maxillary Teeth
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-time i-PRF injection group (Experimental): I-PRF was injected in the buccal region of the mandibular incisors 4 sessions with 28-day interval.
  Interventions: Procedure: 4-time i-PRF injection group
- Control group (Placebo Comparator): Saline serum was injected in the buccal region of the mandibular incisors 4 sessions with 28-day interval
  Interventions: Procedure: Saline injection

INTERVENTIONS:
Procedure: 4-time i-PRF injection group — I-PRF will be injected in 4 sessions at 28-day intervals. The injection will administered submucosally in the buccal region of the lower incisors, using 2 ml of i-PRF per session (0.5 ml per incisor). Orthodontic wires will be sequenced until they reach 0.019×0.025-inch stainless steel.
  Arms: 4-time i-PRF injection group
Procedure: Saline injection — Saline serum will be injected in 4 sessions at 28-day intervals. The injection will be administered submucosally in the buccal region of the lower incisors, using 2 ml of i-PRF per session (0.5 ml per incisor). Orthodontic wires will be sequenced until they reach 0.019×0.025-inch stainless steel.
  Arms: Control group

SUMMARY:
Mandibular incisor crowding is a frequent issue that prompts many adults to seek orthodontic treatment. The treatment may enhance patients' quality of life, facilitate dental plaque control, and improve the quality of periodontal tissue. However, this treatment is accompanied by several side effects, including resorption of the apical portion of the teeth. Platelet-rich concentrates, such as injectable platelet-rich fibrin, have been shown to have positive effects on both soft- and hard-tissue healing. They may serve as a beneficial self-derived material to prevent this complication.

DETAILED DESCRIPTION:
In recent years, increasing attention has been directed toward biologically driven approaches to modulate tissue responses during orthodontic treatment and minimize adverse effects, such as root resorption. Platelet-rich fibrin (PRF), a second-generation autologous platelet concentrate, has emerged as a promising biomaterial due to its high concentration of platelets, leukocytes, and a fibrin matrix that allows gradual release of multiple growth factors, including platelet-derived growth factor (PDGF), transforming growth factor-β (TGF-β), vascular endothelial growth factor (VEGF), and insulin-like growth factor (IGF). However, in 2014, injectable platelet-rich fibrin (I-PRF), which is similar to PRF, was introduced in France by Choukroun, using non-glass tubes and adjusting the centrifugal force. Just like traditional PRF, i-PRF contains high levels of growth factors, stem cells, leukocytes, and cytokines.

These growth factors play a crucial role in angiogenesis, tissue regeneration, modulation of inflammation, and bone remodeling, all of which are central processes in orthodontic tooth movement and periodontal healing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 17 and 28 years
* Class I malocclusion with moderate crowding (4-6 mm) according to Little's Irregularity Index (LII)
* Normal or inclination for mandibular incisors
* Complete permanent teeth.

Exclusion Criteria:

* Previous orthodontic treatment,
* Poor oral hygiene,
* Severe skeletal discrepancy,
* The presence of coagulation disorders or being under anticoagulant treatment.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Change in root length | First assessment time: one day before the commencement of treatment. Second assessment time: within one week following the leveling and alignment stage (The stage is expected to finish within 4 to six months after the beginning of treatment)
  Root resorption (i.e., change in root length) will be measured by calculating the difference in the full linear length of each incisor (incisal edge to the apex) between two assessment times (in millimeters) using CBCT images.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad I. Idris, DDS, Principal Investigator — Faculty of Dentistry, University of Damascus; Ahmad S. Burhan, DDS MSc PhD, Study Director — Faculty of Dentistry, University of Damascus; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Faculty of Dentistry, University of Damascus
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, McGrath C, Hagg U. The impact of malocclusion and its treatment on quality of life: a literature review. Int J Paediatr Dent. 2006 Nov;16(6):381-7. doi: 10.1111/j.1365-263X.2006.00768.x. PMID 17014535
- [Background] Valerio CS, Cardoso CAEA, Araujo EA, Zenobio EG, Manzi FR. Bone changes in the mandibular incisors after orthodontic correction of dental crowding without extraction: A cone-beam computed tomographic evaluation. Imaging Sci Dent. 2021 Jun;51(2):155-165. doi: 10.5624/isd.20200260. Epub 2021 Feb 9. PMID 34235061
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326
- [Background] Samandara A, Papageorgiou SN, Ioannidou-Marathiotou I, Kavvadia-Tsatala S, Papadopoulos MA. Evaluation of orthodontically induced external root resorption following orthodontic treatment using cone beam computed tomography (CBCT): a systematic review and meta-analysis. Eur J Orthod. 2019 Jan 23;41(1):67-79. doi: 10.1093/ejo/cjy027. PMID 29771300
- [Background] Idris MI, Burhan AS, Hajeer MY, Sultan K, Nawaya FR. Efficacy of the injectable platelet-rich fibrin (i-PRF) in gingival phenotype modification: a systematic review and meta-analysis of randomized controlled trials. BMC Oral Health. 2024 Nov 1;24(1):1331. doi: 10.1186/s12903-024-05109-5. PMID 39487452